CLINICAL TRIAL: NCT05642221
Title: Pilot Study of the Use of Functional Near-Infrared Spectroscopy (fNIRS) Combined With Diffuse Correlation Spectroscopy (DCS) in Neurocognitive Disease as Compared to Healthy Neurotypical Controls
Brief Title: Functional Near-Infrared Spectroscopy (fNIRS) Combined With Diffuse Correlation Spectroscopy (DCS) in Neurocognitive Disease as Compared to Healthy Neurotypical Controls
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000862; 000862-CH
Record Dates: First submitted 2022-12-07; First posted 2022-12-08 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-09-29

CONDITIONS: Juvenile Neuronal Ceroid Lipofuscinosis; Smith-Lemli-Opitz Syndrome; Creatine Transporter Deficiency; Niemann-Pick Disease Type C1
Keywords: Brain Hypometabolism; Cerebral Blood Flow; Portable Brain Imaging; Cerebral O2 Changes; Neurocognitive Disorders; Natural History
MeSH Terms: conditions — Neuronal Ceroid-Lipofuscinoses; Smith-Lemli-Opitz Syndrome; Creatine deficiency, X-linked; Niemann-Pick Disease, Type A; Neurocognitive Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: individuals without known health or medical issues (i.e. healthy volunteers)
- 2: individuals with known neurocognitive disorders (i.e. affected)

SUMMARY:
Background:

Neurocognitive disorders affect how the brain uses oxygen. They may affect mental development in children. These disorders can be studied with imaging scans that use radiation; however, these methods are not ideal for research on children. Two technologies-functional near-infrared spectroscopy (fNIRS) and diffuse correlation spectroscopy (DCS)-use light to detect changes in brain activity. These methods are safer, and they can be used in a more relaxed setting. In this natural history study, researchers want to find out whether fNIRS and DCS can be a good way to study people with neurocognitive disorders.

Objective:

To find out whether fNIRS and DCS can be useful in measuring brain activity in people with neurocognitive disorders.

Eligibility:

People aged 6 months or older with neurocognitive disorders. These can include Niemann-Pick disease type C1 (NPC1); creatine transporter deficiency (CTD); Smith Lemli Opitz syndrome (SLOS); juvenile neuronal ceroid lipofuscinosis (CLN3 disease); and Pheland-McDermid (PMS) syndrome. Healthy volunteers are also needed.

Design:

Participants will have a physical exam. They will have tests of their memory and thinking.

Participants will sit in a quiet room for the fNIRS and DCS tests. A snug cap (like a cloth swim cap) will be placed on their head. The cap has lights and sensors. Another sensor will be placed on their forehead. Participants will perform tasks on a computer. This testing will take 45 to 60 minutes.

The tests will be repeated within 1 to 4 weeks. Participants will be asked to return for repeat tests 1 year later.

DETAILED DESCRIPTION:
Study Description:

Brain hypometabolism has been observed in neurologic conditions. These data were obtained using modalities that involved radiation exposure and were not easily amenable to being combined with performance of functional tasks. Functional near-infrared spectroscopy (fNIRS) and Diffusion Correlation Spectroscopy (DCS) are noninvasive, easy-to-use, and portable brain imaging technology that enable studies of metabolic parameters and their alterations with task performance in neurotypical and neurocognitively affected individuals. Specifically, it enables the study of brain oxygen utilization which likely correlates with brain metabolism. We are proposing a pilot study of the use of fNIRS and DCS in neurocognitive disorders that have been extensively followed in our groups: Niemann-Pick disease type C1 (NPC1), creatine transporter deficiency (CTD), Smith Lemli Opitz syndrome (SLOS), Juvenile Neuronal Ceroid Lipofuscinosis (CLN3 disease), and Phelan-McDermid (PMS) syndrome. We want to compare findings in these populations to neurotypical healthy controls.

Objectives:

The primary objective of this pilot study is to determine the feasibility of fNIRS-DCS in individuals with neurocognitive-related disorders.

The secondary objectives of this study are:

1. To collect pilot data on individuals with neurocognitive disorders to determine the patterns of cerebral oxygen consumption as measured by fNIRS and DCS.
2. To compare cerebral oxygen consumption changes from resting state in affected individuals versus age-appropriate healthy volunteers.

An exploratory objective is to correlate cerebral oxygen consumption changes from resting state in affected individuals to other measures of disease state (e.g., neuropsychological assessment, disease-specific severity rating scales). Another exploratory objective is to examine test-retest reliability of our fNIRS-DCS measures at rest and during specific tasks in both affected individuals and healthy controls.

Endpoints:

Primary endpoints:

Adverse events, number of individuals who complete study

Secondary endpoints:

Patterns of cerebral oxygen consumption and blood flow in neurocognitive disorders compared to healthy controls.

ELIGIBILITY:
* INCLUSION CRITERIA:
* For both study populations (Affected and Typically Developing group):

  * Male or female, aged 6 months and up
  * English is the primary language spoken at home
* For study population (Affected group):

  --Neurocognitive-related conditions including SLOS, CLN3, CTD, NPC and PMS.
* For controls (Typically Developing Group):

  * In good general health as determined by medical history and physical exam

EXCLUSION CRITERIA:

* For both study populations (Affected and Typically Developing group):

  * Any condition that may affect placement of the fNIRS-DCS
  * Past or present vascular disease
  * Traumatic loss of consciousness in the last year
  * Any condition which, in the opinion of the investigator, increases risk of participation or affects adherence to the protocol
* For controls (Typically Developing Group):

  * Known or suspected cognitive impairment
  * Known history of MRI abnormality
  * Current use of psychotropic medications

Ages: 6 Months to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: individuals 6 months and older without known health or medical issues (i.e. healthy volunteers), and individuals with known neurocognitive disorders (i.e. affected). Healthy volunteers will be age- and sex-matched to the affected cohort
Sampling Method: Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2025-04-25 (Actual)

PRIMARY OUTCOMES:
Proportion of individuals who complete the study relative to those in which data collection was attempted | 2 years
  We hypothesize that fNIRS and DCS will show low rates of adverse events across all participants (<5%) and high rates of completed fNIRS-DCS data collections (> 75%).
Adverse events | 2 years
  We hypothesize that fNIRS and DCS will show low rates of adverse events across all participants (<5%) and high rates of completed fNIRS-DCS data collections (> 75%).

SECONDARY OUTCOMES:
Cerebral activation, measured via O2 changes, in resting and in active state | 2 years
  We hypothesize that fNIRS and DCS will show cerebral oxygen consumption differences between neurocognitive disorders and age-matched typically developing controls.
Cerebral blood flow in resting and active state | 2 years
  We hypothesize that fNIRS and DCS will show cerebral oxygen consumption differences between neurocognitive disorders and age-matched typically developing controls.

CONTACTS AND LOCATIONS:
Overall Officials: Forbes D Porter, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000862-CH.html